CLINICAL TRIAL: NCT01787812
Title: California Joint Replacement Registry
Acronym: CJRR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: California Joint Replacement Registry (Network)
Responsible Party: Sponsor
Other Study IDs: CJRR-2013
Record Dates: First submitted 2013-02-01; First posted 2013-02-11 (Estimated); Last update posted 2013-07-04 (Estimated); Status verified 2013-07

CONDITIONS: Hip and Knee Replacement Surgeries

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No

SUMMARY:
The California Joint Replacement Registry (CJRR) was created to meet the need for comprehensive, scientific assessment of devices, treatment protocols, surgical approaches, and patient factors influencing the results of hip and knee replacement surgeries. Importantly, it is a Level 3 registry, meaning it collects and incorporates clinical information and direct feedback from patients about the outcomes of hip and knee replacement surgeries. It is one of only a small number of registries in the United States to do so.

The CJRR's goals are to:

* Collect and report scientifically valid data on the results of hip and knee replacements performed in California, including device safety and effectiveness, post-operative complication and revision rates, and patient-reported outcomes; and
* Promote the use of performance information regarding hip and knee replacements to guide physician and patient decisions and to support programs for provider recognition and reward.

Specifically the CJRR is designed to:

* Minimize burden on participants by using electronic data sources, rather than manual data entry or chart review.
* Compile reports assessing the outcomes associated with different devices and surgical techniques.
* Create benchmarking reports for physicians and hospitals that detail performance data and compare it to statewide averages.
* Transmit safety alerts on devices with short-term results that provoke concern.
* Shape a measurement and reporting system for total hip and total knee replacement surgeries.

The CJRR was developed by the California HealthCare Foundation (CHCF), the Pacific Business Group on Health (PBGH), and the California Orthopaedic Association (COA). PBGH manages the day-to-day operations of the CJRR.

CJRR's data elements are aligned with other major orthopedic registries. The CJRR is a member of the International Consortium of Orthopedic Registries (ICOR) and the International Society of Arthroscopic Registries (ISAR).

ELIGIBILITY:
Inclusion Criteria:

* Receiving hip or knee replacement surgery in California.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Californians, 18+ years of age, receiving hip or knee replacement surgery in California.
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2011-07; Primary Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Number of Patients with Total Hip Replacement | 3 months, 6 months, every year up to 5 years
Number of Patients with Partial Hip Replacement | 3 months, 6 months, every year up to 5 years
Number of Patients with Hip Revision | 3 months, 6 months, every year up to 5 years
Number of Patients with Total Knee Replacement | 3 months, 6 months, every year up to 5 years
Number of Patients with Knee Revision | 3 months, 6 months, every year up to 5 years

SECONDARY OUTCOMES:
Number and Type of Adverse Events as a Measure of Patient Safety | 3 months
  Adverse Events:
  * Would infection
  * Fracture
  * Excessive bleeding
  * DVT proximal
  * DVT
  * PE
  * Congestive heart
  * Arrhythmia
  * Renal failure
  * Nerve injury
  * MI
Number and Type of Readmissions as a Measure of Surgical Quality | 3 months, 6 months, every year up to 5 years
Number of Revisions as a Measure of Surgical Quality | 3 months, 6 months, every year up to 5 years
Health-Related Quality of Life Score on the SF-12 | 3 months, 6 months, every year up to 5 years
Pain Score on the WOMAC | 3 months, 6 months, every year up to 5 years
Stiffness Score on the WOMAC | 3 months, 6 months, every year up to 5 years
Physical Function Score on the WOMAC | 3 months, 6 months, every year up to 5 years
Activity Level Score on the UCLA Activity Index | 3 months, 6 months, every year up to 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Hoag Orthopedic Institute, Irvine, California, United States